CLINICAL TRIAL: NCT00603265
Title: A Phase 2a, Randomized, Double-Blind, Placebo- and Active-Controlled, Parallel-Group, Multicenter Study to Assess the Safety and Efficacy of ADL5859 100 mg BID in Subjects With Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Safety and Efficacy Study of ADL5859 in Participants With Neuropathic Pain Associated With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33CL231
Record Dates: First submitted 2008-01-17; First posted 2008-01-29 (Estimated); Results first posted 2015-07-01 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Peripheral Neuropathy; Neuropathic Pain
Keywords: Diabetic Peripheral Neuropathy; Neuropathic Pain
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia | interventions — N,N-diethyl-4-(5-hydroxyspiro(chromene-2,4'-piperidine)-4-yl)benzamide; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ADL5859 (Experimental): 2 x 50 milligrams (mg) ADL5859 capsules administered orally once in the morning and once in the evening for 28 days
  Interventions: Drug: ADL5859
- Duloxetine (Active Comparator): 2 x 30 mg duloxetine capsules administered orally once in the morning and 2 placebo capsules filled with lactose administered orally once in the evening for 28 days
  Interventions: Drug: Duloxetine; Drug: Placebo
- Placebo (Placebo Comparator): 2 placebo capsules filled with lactose administered orally once in the morning and once in the evening for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ADL5859
  Arms: ADL5859
Drug: Duloxetine
  Other Names: Cymbalta
  Arms: Duloxetine
Drug: Placebo
  Arms: Duloxetine; Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of ADL5859 in relieving the pain associated with diabetic peripheral neuropathy (DPN) compared with placebo and duloxetine (a marketed drug approved for the treatment of painful DPN). The pain symptoms of DPN are thought to be due to damage to nerves caused by the diabetes.

DETAILED DESCRIPTION:
Participants were permitted to take acetaminophen 650 to 975 mg every 4 to 6 hours (up to a total of 4 grams in 24 hours) as needed for pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between 18 and 75 years of age, inclusive
* Body weight of at least 45 kilograms (kg)
* Diabetes mellitus (type I or II) that is documented to be under stable glycemic control over a period of at least 3 months, as indicated by a glycosylated hemoglobin (HbgAIC) of less than or equal to 12% and a stable dose of insulin or oral diabetic medication for 90 days prior to starting study medication
* No change in diabetic medications is planned for the duration of the study
* Evidence of symmetrical, bilateral pain in the lower extremities due to diabetic peripheral neuropathy (DPN)
* Presence of daily pain due to DPN for at least 3 months
* Score greater than or equal to 3 on the physical examination portion of the Michigan Neuropathy Screening Instrument (MNSI)
* Average weekly pain score of greater than or equal to 4 on the numeric pain rating scale (NPRS) for symmetrical neuropathic pain in the feet and legs
* For male participants, be surgically sterile or agree to use an appropriate method of contraception
* For female participants of childbearing potential, be surgically sterile or using an intrauterine device, or injectable, transdermal, or combination oral contraceptive deemed highly effective by the Food and Drug Administration (FDA)
* Be willing and able to comply with the protocol requirements
* Be able to understand and willing to provide written informed consent in English

Exclusion Criteria:

* Presence of pain conditions that cannot be distinguished from DPN
* Presence of significant renal disease, as indicated by a serum creatinine greater than or equal to 2.0 milligrams per deciliter (mg/dL), or presence of significant hepatic disease
* Have a history of a seizure disorder
* Presence of serious or unstable cardiovascular disease, respiratory disease, hematologic illness, or a psychiatric condition
* History of evidence of symptomatic orthostatic hypotension
* History of a major depressive disorder, generalized anxiety disorder, eating disorder, or substance abuse (including alcohol) within the past year
* History or evidence of mania, bipolar disorder, or psychosis
* History of allergy to acetaminophen or duloxetine
* Score of greater than or equal to 18 on the Beck Depression Inventory II (BDI-II) or score of greater than zero on Item 9 of the BDI-II
* Use of any of the following concomitant medications: fluvoxamine; quinolone antimicrobials (ciprofloxacin and enoxacin); selective serotonin reuptake inhibitors (SSRIs); serotonin norepinephrine reuptake inhibitors (SNRIs); tricyclic antidepressants; opioids; nonsteroidal anti-inflammatory drugs (NSAIDS); anticonvulsants; aspirin (with the exception of low-dose aspirin as cardiovascular prophylaxis); or cytochrome P4503A (CYP3A) and P-glycoprotein transporter inhibitors
* Pregnant, lactating, or plans to become pregnant during the study
* Presence of foot or toe amputation
* Participation in another study with an investigational compound within the previous 30 days prior to study medication administration, or concurrent participation in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Berger, MD, Study Director — Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA)
Locations (27):
- United States (27):
  - Integrated Research Group, Riverside, California
  - Torrance Clinical Research, Torrance, California
  - FPA Clinical Research, Kissimmee, Florida
  - Innovative Research of West Florida, Inc., Largo, Florida
  - Panhandle Family Care Associates & Emerald Coast Research Grp, Inc., Marianna, Florida
  - Renstar Medical Research, Ocala, Florida
  - Radiant Research-St.Petersburg, Pinellas Park, Florida
  - Doctor's Research Network, South Miami, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Laszlo J. Mate, MD, West Palm Beach, Florida
  - The Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Beacon Clinical Research, Brockton, Massachusetts
  - Healthcare Research, Florissant, Missouri
  - Creighton Diabetes Center, Creighton Univ. Sch. of Medicine, Omaha, Nebraska
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Clnical Study Center of Asheville, Asheville, North Carolina
  - Radiant Research-Akron, Mogadore, Ohio
  - Neurology & Neuroscience Center of Ohio, Toledo, Ohio
  - Aquilo Research, Yukon, Oklahoma
  - Clinical Research Consultants, Research Department, Medford, Oregon
  - Advanced Regional Center for Clinical Research (Ankle & Foot Care), Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Nerve & Muscle Center of Texas, Houston, Texas
  - Invisions Consultants LLC, San Antonio, Texas
  - Diabetes & Glandular Disease Research Associates, San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADL5859 | Duloxetine | Placebo
Started | 76 (1 participant was randomized in error and did not receive study medication) | 78 | 72
Received at Least 1 Dose of Study Drug | 75 | 78 | 72
Completed | 69 | 62 | 67
Not Completed | 7 | 16 | 5
Not completed — Adverse Event | 2 | 11 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Lack of Efficacy | 3 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Out of Town, Ran Out of Study Drug | 0 | 1 | 0
Not completed — Participant Left Country, No Responses | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were randomized and treated with study medication.
Groups:
- ADL5859: 2 x 50 mg ADL5859 capsules administered orally once in the morning and once in the evening for 28 days
- Total: Total of all reporting groups
Arm/Group | ADL5859 | Duloxetine | Placebo | Total
Number analyzed (Participants) | 75 | 78 | 72 | 225
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.7 (10.17) | 59.1 (8.71) | 56.2 (8.78) | 58.3 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 39 | 27 | 101
  Male | 40 | 39 | 45 | 124

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Numeric Pain Rating Scale (NPRS) Score
Description: The NPRS is an 11-point scale (0 to 10) with 0 indicating no pain and 10 indicating the worst possible pain. The mean of the daily average scores were calculated from the NPRS pain assessments obtained up to 3 times per day over a 7-day period. Least Squares (LS) means were calculated using analysis of covariance (ANCOVA) with treatment group as a main factor and baseline NPRS score as a covariate. Change from Baseline = NPRS at baseline - NPRS at Week 4; a positive number in the LS mean indicates a reduction in pain intensity from baseline.
Time Frame: Baseline, Week 4
Population: All participants who received at least 1 dose of study medication and had evaluable NPRS data. Baseline-observation-carried-forward (BOCF) was used to impute missing postbaseline values for participants who were discontinued from the study early.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ADL5859 | Duloxetine | Placebo
Number analyzed (Participants) | 75 | 77 | 72
units on a scale | 1.02 (0.225) | 1.74 (0.221) | 1.51 (0.229)

2. Secondary Outcome: Percentage of Responders
Description: A responder was defined as a participant who showed a reduction in average pain (as measured by NPRS) of at least 30% from baseline to Week 4. The NPRS is an 11-point scale (0 to 10) with 0 indicating no pain and 10 indicating the worst possible pain. The percentage of participants who qualified as responders is presented per treatment arm.
Time Frame: Baseline, Week 4
Population: All participants who received at least 1 dose of study medication, completed the 4-week treatment period, and had evaluable NPRS data.
Measure: Number; unit: percentage of participants
Arm/Group | ADL5859 | Duloxetine | Placebo
Number analyzed (Participants) | 69 | 63 | 67
percentage of participants | 26.1 | 52.4 | 38.8

3. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: PGIC is a participant-rated instrument that measures the change in the participant's overall status for the previous 2 weeks based on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). The number of participants in each category is presented.
Time Frame: Week 4
Population: All participants who received at least 1 dose of study medication, completed the 4-week treatment period, and had evaluable PGIC data.
Measure: Number; unit: participants
Arm/Group | ADL5859 | Duloxetine | Placebo
Number analyzed (Participants) | 69 | 63 | 67
participants
  Very Much Improved | 7 | 11 | 11
  Much Improved | 20 | 15 | 11
  Minimally Improved | 20 | 17 | 22
  No Change | 19 | 14 | 21
  Minimally Worse | 0 | 2 | 0
  Much Worse | 3 | 1 | 1
  Very Much Worse | 0 | 1 | 0
  Not Reported | 0 | 2 | 1

4. Secondary Outcome: Change in Sleep Interference Scale (SIS) From Baseline
Description: Sleep Interference was assessed on an 11-point Numeric Rating Scale where a score of 0 indicated "pain did not interfere with sleep" and a score of 10 indicated "pain completely interfered with sleep". Here, "n" signifies "Number of participants" for Baseline and Month 3 telephone interview whereas "n" signifies "number of observations" for Month 1, 2, and 3 because a participant could have had multiple visits during Month 1, 2, and 3 as this was a non-interventional study with no scheduled study visits, except Baseline visit and the Month 3 telephone interview. LS means were calculated using ANCOVA with treatment group as a main factor and baseline SIS score as a covariate. Change from baseline = SIS score at baseline - SIS score at Week 4.
Time Frame: Baseline, Week 4
Population: All participants who received at least 1 dose of study medication, completed the 4-week treatment period, and had evaluable SIS data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ADL5859 | Duloxetine | Placebo
Number analyzed (Participants) | 69 | 63 | 66
units on a scale | 1.92 (0.291) | 2.27 (0.304) | 1.56 (0.297)

5. Secondary Outcome: Change From Baseline in the Evening Assessment of the 24-hour Overall Mean Pain Intensity Score
Description: At each of the evening pain assessments, participants assessed their overall pain intensity over the preceding 24 hours using NPRS. The NPRS is an 11-point scale (0 to 10) with 0 indicating no pain and 10 indicating the worst possible pain. The mean of the daily average scores were calculated from the NPRS pain assessments obtained at Baseline and Week 4. Change from baseline = NPRS at baseline - NPRS at Week 4.
Time Frame: Baseline, Week 4
Population: All participants who received at least 1 dose of study medication and had evaluable 24-hour NPRS data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADL5859 | Duloxetine | Placebo
Number analyzed (Participants) | 69 | 63 | 67
units on a scale | 1.09 (1.847) | 2.15 (2.322) | 1.51 (2.027)

6. Secondary Outcome: Change From Baseline in NPRS at Rest in the Clinic
Description: The mean of the daily average scores were calculated from the NPRS pain assessments obtained 1 time per week over a 4-week period. NPRS assessments were taken while the participant was at rest. The NPRS is an 11-point scale (0 to 10) with 0 indicating no pain and 10 indicating the worst possible pain. LS means were calculated using ANCOVA with treatment group as a main factor and baseline NPRS score as a covariate. Change from baseline = NPRS at baseline - NPRS at Weeks 1, 2, 3, and 4.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: All participants who received at least 1 dose of study medication, completed the 4-week treatment period, and had evaluable at-rest NPRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ADL5859 | Duloxetine | Placebo
Number analyzed (Participants) | 69 | 63 | 67
units on a scale
  Week 1 (n=67, 59, 64) | 0.70 (0.200) | 1.15 (0.213) | 0.75 (0.205)
  Week 2 (n=68, 61, 65) | 0.80 (0.237) | 1.44 (0.250) | 1.16 (0.243)
  Week 3 (n=67, 61, 63) | 0.92 (0.265) | 1.95 (0.277) | 1.27 (0.274)
  Week 4 (n=68, 61, 65) | 1.13 (0.269) | 2.03 (0.283) | 1.59 (0.276)

7. Secondary Outcome: Change From Baseline in NPRS After Walking 50 Feet in the Clinic
Description: The mean of the daily average scores were calculated from the NPRS pain assessments obtained 1 time per week over a 4-week period. NPRS assessments were taken after the participant walked 50 feet in the clinic. The NPRS is an 11-point scale (0 to 10) with 0 indicating no pain and 10 indicating the worst possible pain. LS means were calculated using ANCOVA with treatment group as a main factor and baseline NPRS score as a covariate. Change from baseline = NPRS at baseline - NPRS at Weeks 1, 2, 3, and 4.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4
Population: All participants who received at least 1 dose of study medication, completed the 4-week treatment period, and had evaluable post-walk NPRS data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ADL5859 | Duloxetine | Placebo
Number analyzed (Participants) | 69 | 63 | 67
units on a scale
  Week 1 (n=67, 59, 64) | 0.88 (0.215) | 1.42 (0.229) | 1.00 (0.220)
  Week 2 (n=67, 61, 65) | 0.93 (0.254) | 1.75 (0.267) | 1.23 (0.259)
  Week 3 (n=67, 61, 63) | 1.24 (0.281) | 2.25 (0.294) | 1.43 (0.290)
  Week 4 (n=68, 61, 65) | 1.29 (0.273) | 2.36 (0.288) | 1.79 (0.279)

ADVERSE EVENTS:
Groups:
- Duloxetine: 2 placebo capsules filled with lactose administered orally once in the morning and once in the evening for 28 days
- Placebo: 2 x 30 mg duloxetine capsules administered orally once in the morning and 2 placebo capsules filled with lactose administered orally once in the evening for 28 days
Arm/Group | ADL5859 | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/75 | 1/78 | 0/72
Other Adverse Events (participants affected / at risk) | 27/75 | 28/78 | 27/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADL5859 (N=75) | Duloxetine (N=78) | Placebo (N=72)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 — Resulted in one death in the duloxetine group.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ADL5859 (N=75) | Duloxetine (N=78) | Placebo (N=72)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Bundle branch block (Cardiac disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 1 | 2 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 9 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Dysgeusia (Gastrointestinal disorders) | 0 | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 16 | 3
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0
Asthenia (General disorders) | 1 | 3 | 1
Fatigue (General disorders) | 1 | 3 | 3
Feeling hot (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 2
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 3
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 2
Viral infection (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1/35 | 0/39 | 0/27
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 1 | 1
Blood potassium increased (Investigations) | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1
Eosinophil count increased (Investigations) | 3 | 0 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 5 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 1
Essential tremor (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 6 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 3 | 0
Tremor (Nervous system disorders) | 0 | 3 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Libido decreased (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0/35 | 0/39 | 1/27
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 7 | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other